CLINICAL TRIAL: NCT02373878
Title: Telecoaching Plus a Portion Control Device for Weight Care Management
Brief Title: Telecoaching Plus a Portion Control Device for Weight Management in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jon Ebbert, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11001395
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telecoaching plus plate (Active Comparator): Telecoaching plus portion control plate
  Interventions: Behavioral: Telecoaching plus Plate
- Usual Care (Active Comparator): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telecoaching plus Plate — A wellness coach proactively contacted the participants every two weeks during treatment, using motivational interviewing. In addition, she provided a portion control plate.
  Arms: Telecoaching plus plate
Behavioral: Usual Care — Subjects were provided with institutional pamphlets on healthy eating and exercise habits
  Arms: Usual Care

SUMMARY:
The purpose of this study was to evaluate the impact of telecoaching conducted by a counselor trained in motivational interviewing paired with a portion control device for obese patients receiving care in a certified patient-centered medical home. The investigators will conduct a randomized, controlled clinical trial evaluating the effectiveness of a telecoaching intervention with a portion control device.

DETAILED DESCRIPTION:
The intervention will be provided during a 3-month period with follow-up through 6 months after randomization. Body mass index (BMI) and waist circumference measurements will be collected at baseline and at 6, 12, 18, and 24 weeks. Participants will also complete measures assessing eating behaviors and physical activity at baseline and at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years and ≤ 55 years of age
* A BMI of ≥ 30 and ≤ 44.9 kg/m2
* Motivated to lose weight
* Able to participate fully in all aspects of the study;
* Have been provided with, understand, and have signed the informed consent.

Exclusion Criteria:

* Unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months or an untreated cardiac dysrhythmia
* A history of a gastric bypass procedure or planned gastric bypass
* Baseline systolic blood pressure > 180 or diastolic > 100
* Another member of their household already participating in this study
* Current treatment with another investigational drug for obesity (within 30 days of study entry)
* Are pregnant or lactating
* History of anorexia or bulimia
* Current binge eating disorder as assessed by the Patient Health Questionnaire eating disorder module (PHQ-ED)
* Schizophrenia or bipolar disorder or have a PHQ-2 ≥ 337
* Have been diagnosed with cancer within the past 5 years
* Are currently participating in a program specifically to lose weight or are on a weight loss medication (last 30 days)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon O Ebbert, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Huber JM, Shapiro JS, Wieland ML, Croghan IT, Vickers Douglas KS, Schroeder DR, Hathaway JC, Ebbert JO. Telecoaching plus a portion control plate for weight care management: a randomized trial. Trials. 2015 Jul 30;16:323. doi: 10.1186/s13063-015-0880-1. PMID 26223309